CLINICAL TRIAL: NCT04970433
Title: The Effects of Electroacupuncture and Laser Acupuncture Therapy for Patients With Major Trauma
Brief Title: The Effects of Acupuncture for Major Trauma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMRPG8L6041
Record Dates: First submitted 2021-07-12; First posted 2021-07-21 (Actual); Last update posted 2022-03-31 (Actual); Status verified 2021-07

CONDITIONS: Major Trauma
Keywords: major trauma; acupuncture; laser acupuncture
MeSH Terms: interventions — Electroacupuncture

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Electroacupuncture (EA) (Experimental): Acupoint regimen: Hegu (LI4), Neiguan (PC6), Zusanli (ST36), Sanyinjiao (SP6) and Sishencong (EX-HN1). Electrical stimulation using an EA apparatus, with a pair of electrodes connecting acupoints LI4 with PC6, and another pair of electrodes connecting ST36 with SP6. EA stimulation will last for 15 min with a continuous wave of 2 Hz and a current intensity of 0.1-1 mA.
  Interventions: Procedure: Electroacupuncture (EA)
- Laser acupuncture (LA) (Active Comparator): Participants allocated to the LA group will receive LA therapy at the same acupoints used in EA group. The laser will be applied to each point for 40 seconds, which delivered 3 J of energy at each of the acupoints.
  Interventions: Procedure: Laser acupuncture (LA)
- Sham laser acupuncture (SLA) (Sham Comparator): Participants in the control group will receive sham LA treatment without any laser output. The acupuncture points, application duration, and total number of treatments are the same as those in the LA group.
  Interventions: Procedure: Sham laser acupuncture (SLA)

INTERVENTIONS:
Procedure: Electroacupuncture (EA) — Acupuncture at Hegu (LI4), Neiguan (PC6), Zusanli (ST36), Sanyinjiao (SP6) and Sishencong (EX-HN1). Electrical stimulation with a pair of electrodes connecting on LI4/PC6 and ST36/SP6.
  Arms: Electroacupuncture (EA)
Procedure: Laser acupuncture (LA) — The laser applies to each point for 40 seconds, which delivers 3 J of energy at each of the acupoints as those in electroacupuncture group.
  Arms: Laser acupuncture (LA)
Procedure: Sham laser acupuncture (SLA) — The laser device without any laser output applies on the acupoints the same as those in the LA group.
  Arms: Sham laser acupuncture (SLA)

SUMMARY:
Major trauma is a significant cause for morbidity and mortality in the world. After traumatic injury, the damage tissue could induce systemic inflammatory response (SIRS) and activate autonomic nervous system in response to stress, followed by compensatory anti-inflammatory response (CARS). Imbalance of SIRS and CARS may lead to organ failures, sepsis and death.

DETAILED DESCRIPTION:
The investigators design a prospective clinical trial to investigate the efficacy of acupuncture for major trauma.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 20 years or older
* Confirmed diagnosis of major trauma with ISS ≥ 16

Exclusion Criteria:

* Pregnancy
* Malignancy
* Pacemaker
* Status epilepticus
* Severe medical disease
* Life threatening
* Prior history of drug or alcohol dependence
* Immunodeficiency
* Vagotomy

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 180 (Estimated)
Dates: Start 2021-10-12 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-07 (Estimated)

PRIMARY OUTCOMES:
Length of hospital stay | up to 24 weeks
  Count the total days of hospitalization

SECONDARY OUTCOMES:
CRP | measured at 48 hours, 7 days and 14 days
  Inflammatory mediator, CRP
IL-6 | measured at 48 hours, 7 days and 14 days
  Inflammatory mediator, IL-6
TNF-α | measured at 48 hours, 7 days and 14 days
  Inflammatory mediator, TNF-α
IL-1β | measured at 48 hours, 7 days and 14 days
  Inflammatory mediator, IL-1β
IL-10 | measured at 48 hours, 7 days and 14 days
  Inflammatory mediator, IL-10
Sequential organ failure assessment (SOFA) score | measured at 48 hours, 7 days and 14 days
  The SOFA score is a simple and objective score that allows for calculation of both the number and the severity of organ dysfunction in six organ systems (respiratory, coagulatory, liver, cardiovascular, renal, and neurologic), and the score can measure individual or aggregate organ dysfunction.The SOFA score ranges from 0 to 24; higher scores mean a worse outcome.
WHO Disability Assessment Schedule 2.0 (WHODAS 2.0) 12-item version | measured at 3 and 6 months
  WHODAS 2.0 is used to measure of disability after major trauma.
Peripheral Blood Mononuclear Cell (PBMC) analysis | measured at 48 hours, 7 days and 14 days
  PBMC analysis by flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Chun-Ting Liu, Dr., Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Kaohsiung Chang Gung Memorial Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: No
For patient privacy and research confidentiality, temporarily not open.

REFERENCES:
- [Derived] Liu CT, Hsieh TM, Shih FY, Lai WH, Hsieh CH, Wu BY, Chen YH. The effects of electroacupuncture and laser acupuncture therapy for patients with major trauma: A study protocol. Medicine (Baltimore). 2021 Dec 30;100(52):e28367. doi: 10.1097/MD.0000000000028367. PMID 34967368